CLINICAL TRIAL: NCT07217067
Title: A Randomized, Placebo-controlled, Participant- and Investigator-blinded Study to Evaluate the Efficacy in Reducing Atrial Fibrillation Burden (AFB) as Well as the Safety, Tolerability, and Pharmacokinetics of Oral PKN605 in Participants With Atrial Fibrillation
Brief Title: A Study to Investigate the Efficacy, Safety, Tolerability and Pharmacokinetics of PKN605 in Participants With Atrial Fibrillation
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CPKN605A12201
Record Dates: First submitted 2025-10-14; First posted 2025-10-15 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Atrial Fibrillation
Keywords: Atrial fibrillation; Atrial fibrillation burden; Arrythmia
MeSH Terms: conditions — Atrial Fibrillation; Arrhythmias, Cardiac

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- PKN605 lower dose (Experimental): PKN605 is an oral fomulation
  Interventions: Drug: PKN605
- PKN605 higher dose (Experimental): PKN605 is an oral formulation
  Interventions: Drug: PKN605
- Placebo (Placebo Comparator): Placebo is an oral formulation
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: PKN605 — PKN605 is an oral formulation
  Arms: PKN605 higher dose; PKN605 lower dose
Other: Placebo — Matching placebo
  Arms: Placebo

SUMMARY:
A randomized, placebo-controlled, participant-and investigator-blinded study to evaluate the efficacy in reducing atrial fibrillation burden as well as the safety, tolerability and pharmacokinetics of PKN605 in participants with atrial fibrillation

DETAILED DESCRIPTION:
A screening period of up to 90 days will be conducted to determine participants' eligibility. Once eligibility is confirmed, participants will be randomly assigned to receive either PKN605 or placebo. The treatment phase will last for 24 weeks, during which participants will visit the clinic approximately once a month. During the study, participants' atrial fibrillation will be monitored using various ECG devices. Approximately one month after the end of the treatment phase, participants will have a final safety follow-up visit. The primary purpose of the study is to monitor the effect PKN605 has on the amount of time participants spend in atrial fibrillation.

ELIGIBILITY:
Inclusion Criteria:

* Inclusions at Screening

  * Signed informed consent must be obtained prior to participation in the study
  * Male and female participants ≥ 18 years of age
  * History of at least 2 episodes of AF
  * At least 1 of the AF episodes specified in inclusion #3 must be within the last 12 months (or during screening) and documented by 12-lead ECG, Holter, or any other ECG recording method, as confirmed by the Investigator
  * One or more of the following:
* AFB of 1% or higher on a local ambulatory Holter, mobile cardiac telemetry, ECG patch monitor, or other ambulatory electrocardiographic monitor within the last 12 months
* CHA2DS2-VASc score of 2 or higher in males, 3 or higher in females (1 point for congestive heart failure, hypertension, age 65-74 years, diabetes, vascular disease, female sex; 2 points for age 75 years or older, prior stroke or transient ischemic attack)
* Stable heart failure or with New York Heart Association class I or II symptoms
* NT-proBNP level of 300 pg/mL or higher on a local lab test within the last 12 months

  * On guideline-directed stroke prevention treatment, as confirmed by the Investigator
  * Participants must have a body mass index (BMI) ≥ 18 kg/m2. BMI is calculated as body weight (kg) divided by height (m) squared
* Inclusions at Day 1

  * Sinus rhythm at Baseline documented by 12-lead ECG (participants with persistent AF should be cardioverted at least 12 hours before randomization)

Exclusion Criteria:

-Exclusions at Screening

* Permanent AF
* Ongoing reversible causes of AF (e.g., hyperthyroidism, myocarditis, acute alcohol, sepsis- or infection related AF, surgery-related AF, pulmonary embolism)
* Ongoing use of antiarrhythmic therapy (Vaughan Williams class I or III anti-arrhythmic therapy must be discontinued at least 7 days before Screening phase ECG patch monitor; amiodarone must be discontinued at least 6 weeks before Screening phase ECG patch monitor)
* History of an AF ablation procedure within the last 6 months without a recurrence of AF at least 2 or more months after the ablation.
* Implanted pacemaker, defibrillator, or cardiac monitor
* Infiltrative (e.g., amyloidosis, sarcoidosis) or hypertrophic cardiomyopathy
* Left ventricular ejection fraction of 40% or less documented within the last 12 months, or during Screening
* Current decompensated heart failure or hospitalization for heart failure within 3 months prior to Screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 165 (Estimated)
Dates: Start 2025-10-28 (Actual); Primary Completion 2027-09-09 (Estimated); Study Completion 2027-09-09 (Estimated)

PRIMARY OUTCOMES:
Atrial fibrillation burden from ECG patch monitors | 24 weeks
  Defined as the amount of time spent in atrial fibrillation as a proportion of the analyzable monitoring time

SECONDARY OUTCOMES:
Time from the date of randomization to first atrial fibrillation recurrence | 24 weeks
  Defined as the time (days) from the date of randomization to first atrial fibrillation recurrence
Presence of atrial fibrillation recurrence after randomization | 24 weeks
  Defined as presence of (or absense) of atrial fibrillation recurrence after randomization detected by ECG patch monitor, 12-lead ECG, handheld ECG, or other protocol approved method for ascertainment individually and as a composite
Pharmacokinetic Parameter: concentration | 24 Weeks ( 0 hour(Pre-dose), 2 and 4 hour post dose)
  PKN605 plasma concentration

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (22):
- United States (4):
  - Cardiology Associates of North MS, Tupelo, Mississippi
  - Weill Cornell Medical Center, New York, New York
  - Intermountain Medical Center, Murray, Utah
  - Swedish Heart and Vascular Clinic, Seattle, Washington
- Canada (6):
  - Novartis Investigative Site, London, Ontario
  - Novartis Investigative Site, Newmarket, Ontario
  - Novartis Investigative Site, Toronto, Ontario
  - Novartis Investigative Site, Montreal, Quebec
  - Novartis Investigative Site, Québec, Quebec
  - Novartis Investigative Site, Sherbrooke, Quebec
- China (2):
  - Novartis Investigative Site, Beijing, Beijing Municipality
  - Novartis Investigative Site, Xi'an
- Germany (3):
  - Novartis Investigative Site, Bad Homburg
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Hamburg
- Netherlands (3):
  - Novartis Investigative Site, Delft, South Holland
  - Novartis Investigative Site, Goes, Zeeland
  - Novartis Investigative Site, Veldhoven
- Singapore (2):
  - Novartis Investigative Site, Singapore, Singapore
  - Novartis Investigative Site, Singapore
- United Kingdom (2):
  - Novartis Investigative Site, Brighton, East Sussex
  - Novartis Investigative Site, London

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com